CLINICAL TRIAL: NCT02394197
Title: Comparison of the Effectiveness of Two Scheme Treatments to Treat Plasmodium Vivax Cases in Patients Living in Communities With Persistence of Transmission in Oaxaca and Chiapas, Mexico
Brief Title: Effectiveness of Malaria Treatment in Mexico
Acronym: EMTM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LILIA GONZALEZ CERON (Other)
Collaborators: Instituto de Diagnóstico y Referencia Epidemiológicos (InDRE), Mexico (Unknown); Centro Nacional de Vigilancia Epidemiológica y control de enfermedades (CENAVECE), Mexico (Unknown); Jurisdicción Sanitaria VII, Chiapas, México (Unknown); Pan American Health Organization (Other)
Responsible Party: Sponsor-Investigator, LILIA GONZALEZ CERON, Researcher in medical Sciences, Instituto Nacional de Salud Publica, Mexico
Organization: Instituto Nacional de Salud Publica, Mexico (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INSP CI-624; PAHO-MEX/07/005015 (Other Grant/Funding Number: Pan American Health Organization); PAHOERC-162-MEX (Registry Identifier: Pan American Health Organization)
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Malaria
Keywords: Plasmodium vivax; Mexico; treatment; chloroquine; primaquine; 14-day treatment (T14); intermittent single doses (ISD)
MeSH Terms: conditions — Malaria; Malaria, Vivax | interventions — chloroquine diphosphate; Chloroquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 14-day treatment (T14) (Active Comparator): The operational treatment-dose was administered by mouth. The number of tablets of Chloroquine phosphate of 150 mg for three days (x-x-x/ number of tablets of Primaquine (15mg or 5 mg)), daily during 14 days. For 1 year old subjects only chloroquine (1-½-½/ ½ of 5 mg); for 2-5 years old (1-¾-1/ 1 of 5 mg); 6-12 years old (2-1-2/ 2 of 5 mg); 13 years old and over with about 60 kg of body weight (3-2-2/ 1 of 15 mg) and above 60 kg of body weight (4-3-3 / 1 of 15 mg).
  According to the age group as indicated by the Mexican guidelines for vector borne diseases control (http://www.salud.gob.mx/unidades/cdi/nom/032ssa202.html) (Table 10)
  Interventions: Drug: Chloroquine phosphate; Drug: primaquine
- Intermittent single doses (ISD) (Experimental): The single dose medication was administered orally according to age group as the operational table: (number of tablets of chloroquine phosphate of 150 mg / number of tablets of primaquine (15mg or 5 mg)): for 1 year old (½ / 1 of 5 mg); for 2¬-5 years old (1 / 2 of 5 mg); 6-12 years old (2 / 4 of 5 mg); 13 years old and over of about 60 kg of body weight (3 / 2 of 15 mg), and above 60 kg of body weight (4 / 3 of 15 mg).
  It is administered on Days 0 (after the detection of infection by microscopy), and Days 30, 60, 180, 210, 240 and 360 as indicated in the National guidelines for vector borne diseases control (http://www.salud.gob.mx/unidades/cdi/nom/032ssa202.html).
  Interventions: Drug: Chloroquine phosphate; Drug: primaquine

INTERVENTIONS:
Drug: Chloroquine phosphate — use at operational doses by age group according to the Mexican guidelines for vector borne diseases
  Other Names: aralen
Drug: primaquine — use at operational doses by age group according to the Mexican guidelines for vector borne diseases

SUMMARY:
In the context of malaria elimination in the Americas, solid evidence is necessary of the effectiveness of anti-malarial control measures delivered to the affected individuals. In the Americas, most P. vivax infections are sensitive to Chloroquine (CQ) and Primaquine (PQ), and the most effective treatment worldwide comprises administration of a total dose of 25 milligrams (mg)/Kilogram (kg) weight of CQ distributed in three days and 3.5 mg/kg body weight of PQ administered during 14 days (T14). In Mexico, CQ and PQ have been administered since the late 50´s to treat malarious patients. In 1999 the National Malaria Control Program implemented an intermittent single doses treatment (ISD) as part of the overall strategy. After the blood sample was obtained for diagnosis of symptomatic patients, a single combined dose of CQ and PQ was administered, and after malaria infection confirmation, additional doses were administered monthly alternating each three months, during 3 years. Although, the number of malaria cases were reduced in most affected regions, in Southern México, many patients under ISD present recurrent blood infections, presumably relapse episodes were observed.

Working hypothesis: the administration of ISD is low effective to eliminate relapse episodes and its effectiveness depends on the coincidence of the relapse episodes and the administration of the medication), while the T14 is highly effective to eliminate P. vivax primary and relapse infections.

Objective: To determine the antimalarial drug effectiveness of the ISD and T14, based on CQ and PQ for the treatment of uncomplicated P. vivax infection (primary and recurrent blood infections) in Southern Mexico.

Methods: The study was carried out in malaria affected communities of Southern Mexico, following the WHO recommendations for clinical studies. Symptomatic patients diagnosed with P. vivax infection that meet the inclusion criteria, were invited to participate. After they accepted by informed consent, patients were semi-randomized and treated with either T14 (14-day treatment) or ISD (18 intermittent single doses of CQ-PQ). Clinical, parasitological, molecular and serological parameters were monitor over a 12-month follow up period to evaluate the treatment outcomes to cure blood infection and relapsing episodes. The study was conducted from February-2007 to October-2010. The results of this study will be used to assist the Ministry of Health of México in assessing the current national treatment guidelines for uncomplicated P. vivax malaria

DETAILED DESCRIPTION:
Malaria is in pre-elimination status in Mexico (Rodriguez et al., 2011; WHO, 2012) the local transmission of Plasmodium falciparum was interrupted since 2000, and transmission of P. vivax, the only causative agent in the country, is reduced to very few hot spots (Ministry of Health - Mexico, 1995-2005, Pan American Health Organization (PAHO), 2008, WHO, 2012).

Cloroquine (CQ) and primaquine (PQ) are used since 1940 to treat P. vivax blood and liver infections in most affected areas worldwide (Coatney, 1963). However P. vivax resistant to CQ has been progressively reported in various geographic regions since the late 80´s, (Baird 1995). Chloroquine, no longer recommended as mono-therapy WHO, 2010), administered (25 mg / Kg. body weight) during three consecutive days (10,10 and 5 mg /Kg body weight) in combination with PQ (0.25 - 0.75 mg/Kg body weight) during 14 days, is still used in regions were parasites are susceptible (White, 1998; WHO, 2010). The 14 -day regimen effectively cures primary blood infections and prevents relapses in at least 90% of patients (Galappaththy et al., 2007).

In Mexico, CQ combined with PQ has been used as the standard treatment for P. vivax malaria since the 50´s of the past century. However, PQ treatment is frequently not completed due to undesirable side effects such as stomach upsetting. In locations of difficult access, the extended intervals between blood sampling, parasitological diagnosis and treatment of patients could take as long as 3-4 weeks. Hence, to reduce the risk of transmission, febrile patients in remote areas were blood sampled and immediately treated with a single dose of 10 mg CQ and 0.75 mg PQ/kg body weight, and, only after microscopy confirmation, an intermittent single dose regimen (ISD) was administered (Mendez et al., 1994; Channon et al., 2003; NOM-032-SSA2-2002).

The first single combined CQ-PQ is still administered and it is expected to eliminate blood parasites since PQ may destroy parasites surviving from the effect of CQ [Murphy et al., 1991), and the repeated administration of ISD was intended to suppress parasitemia recurrences (Mendez et al., 1994). However, its effectiveness has not been evaluated.

Assessment and monitoring of the effectiveness of the implemented treatment strategies are necessary to advance towards malaria elimination in the region (malERA, 2011).

Methodology This study was approved by the Ethical Review Committee of the National Institute of Public Health (INSP), Mexico. Informed consent was obtained from all patients and the guardians of patients under 18 years old.

The study followed the World Health Organization (WHO) in vivo test protocol for monitoring antimalarial drug resistance. Since early relapses can occur after 17 days post-primary blood infection, for the primary blood infection clearance, patients were followed up for ≈Day 28 and from one month and up to 12 months to monitor relapse elimination. When required, a flexible schedule was implemented to facilitate patients' follow up and minimized patient lost as suggested by others (Ruebush et al., 2003).

Study site. The study was carried out in Tapachula municipality and surrounding communities in southern Chiapas, Mexico, bordering Guatemala. Patient recruitment was carried out in the diagnosis facility at the Regional Center for Public Health Research-INSP (CRISP) in Tapachula City, where febrile people seeking malaria diagnosis and treatment, obtain free services.

Sample size. A minimum sample size of participants per group was expected as indicated by The World Health Organization for clinical studies in the Americas ((WHO, 2009; PAHO, 2010). However, the total patients enrolled during the study period, was determined by the number of cases diagnosed with P. vivax that meet the inclusion criteria and accepted to participate.

Patient enrollment. A symptomatic patient was defined as a person that presented fever or two other malaria symptoms. Patients were recruited from February 2008 to October 2009 following the inclusion and exclusion criteria (see eligibility criteria). Enrolled patients were randomized to receive either, combined CQ and PQ medication in ISD or T14 schemes, but patients living in Tapachula City and nearby were preferred to receive T14 to facilitate daily treatment supervision. The same day of diagnosis and prior treatment administration (day 0; date annotated), patients were examined for axial temperature in celsius degree (°C), body weight (in kg), spleen swelling and the presence of clinical symptoms within the previous 48 h as fever, headache, myalgia and arthralgia. Erythema and jaundice signs were determined at day of enrollment. For parasitological and molecular analysis, Capillary blood was collected by finger pricking to prepare thin and thick smears and to impregnate filter papers (Whatman #2), respectively. Other demographic data were collected using a questionnaire e.g. age, gender, previous chloroquine and primaquine intake and malaria infections, etc.

Patient treatment and follow-up. The recommended dose for one single dose consisted of 10 mg/kg of CQ phosphate and 0.75 mg/kg of primaquine. Patients under ISD were schedule to take a single dose on Days 0, 30, 60, 180, 210 and 240. On the other hand, the optimal dose of T14 included 25 mg/kg of CQ administered over a 3-day period (10 mg/kg on days 0 and 1 and 5 mg/kg on day 2) and PQ at 0.25mg/kg/day during 14 days (WHO, 2010). However, both treatment regimens were adjusted to patients' age according to the operational table prescribed by the Mexican official guidelines (NOM-032-SSA2-2002). All treatment doses were administered under the supervision by a member of the study team. For small children, tablets were crushed, mixed with water and spoon fed. Treated patients were observed during 30 minutes after ingesting the drugs. Those who vomited the first dose were re-treated with a similar dose, but those who vomited again were excluded from the study.

The first part of the study was designed to monitor the parasitological (primary blood infection clearance) and clinical responses to both treatment schedules. Treated patients were scheduled for examination on Days 2, 3, 7, 14, 21 and 28. The second part of the study was designed to monitor the occurrence of relapses by monthly parasitological and clinical examinations, up to 12 months.

Patients were encouraged to come back to our facilities, or if necessary to contact us by cell phone (most patients or their parents had a cell phone), if they felt ill at any time during the follow-up period or had any question about the study. Participants unable to return to our facilities were visited at their homes to provide treatment, clinical revision and blood sampling. A rapid diagnostic test (RDT) (OptiMAL©) was applied to symptomatic patients at their homes. The thick smears of symptomatic patients with negative RDT were analyzed the same day and in the case of confirming a recurrent P. vivax episode, patients were immediately treated with T14.

When required, a flexible schedule was implemented to facilitate patients' follow up e.g. if patients after the first SD regimen were not at home on Day 3 they were visited on Day 4, Days 7 ± 1, and Day 14 ± 2, and for all patients (under ISD or T14) on Days 21 ± 2 and so on. Two thick and thin blood films and a sample of blood impregnated in filter paper (Whatman #2) were prepared at every scheduled or extra visit (in symptomatic patients). Patients with axillary temperatures ≥37.5 ◦C were symptomatically treated with paracetamol (10 mg/kg).

(see Outcome measures)

Parasitological diagnosis. Thick and thin blood films were stained with 10% solution of Giemsa colorant for five min. The thick smears were examined under a light microscope using oil immersion 100 × by experienced microscopists. Asexual and sexual parasite densities were determined by counting the number of parasites against 200 white blood cells (WBC) (or 500 WBC, if less than 10 parasites were encountered in 200 WBC fields), assuming 7,000 WBC/μl of blood (Gonzalez-Ceron et al., 2005).

Anti-P. vivax blood stages IgG antibodies by ELISA. To uncover P. vivax recurrent blood infections; asymptomatic and/or of low parasitemia not detected by microscopy, immunoglobulins isotype G (IgG) against native P. vivax blood stage proteins were measured in all samples obtained from month 1 to 12. From each patient, blood samples preserved in filter papers were eluted in phosphate-buffered saline (PBS) and tested in an ELISA to detect IgG antibodies against P. vivax blood stages (Gonzalez-Ceron et al., 1991). Sero-conversion or changes in antibody titers were analyzed. A cut off value of 0.25 of absorbance value was previously determined.

Molecular diagnosis . Molecular diagnosis has been shown to be very sensitive in different malaria affected regions (Rubio et al., 1999). All follow-up blood samples of Days 2, 3, 7, 14, ~21 and ~28, and those samples taken during the 12-month follow up with suspicion of recent malaria infection, suggested by an increase in antibody anti-P. vivax IgG (by ELISA ), were subjected to molecular diagnosis. Six punches of 5 mm of dried blood in filter paper were cut and used to extract DNA using the QIAamp® DNA Blood Mini Kit (QIAGEN, Germany) following the manufacturer instructions. The DNA was suspended in 50 µl of water. To detect the P. vivax RNA ribosomal 18S subunit gene (18ssrRNA).

Genotyping primary and recurrent P. vivax infections (Gonzalez-Ceron et al., 2013). To compare P. vivax genotypes of primary and secondary episodes, Polymerase chain reaction-restriction Fragment Length Polymorphism (PCR-RFLP) was used to analyze cspr, msp3α and msp3β gene markers. The homogeneity of P. vivax genotypes among groups was examined by a Fisher´s exact test (α = 0.05).

Data analysis All parasitological and clinical data from each patient that completed the supervised treatments (for 28 days, and for 12-month) were analyzed using STATA v12. To discard the possibility that a sub-dose caused delay in parasite clearance, the body weights recorded on day 0 was used to calculate doses of CQ and PQ given to patients and compared to that necessary for their body weight.

Parasitological and clinical cure of the primary blood infection:

Classification of treatment outcomes as indicated by the methods of surveillance of antimalarial drug efficacy (WHO, 2009)

Early treatment failure (ETF)

* danger signs or severe malaria on day 1, 2 or 3 in the presence of parasitaemia;
* parasitaemia on day 2 higher than on day 0, irrespective of axillary temperature;
* parasitaemia on day 3 with axillary temperature ≥ 37.5 ºC;
* parasitaemia on day 3 ≥ 25% of count on day 0. Late treatment failure (LTF)
* Danger signs or severe malaria in the presence of parasitaemia on any day between day 4 and day 28 in patients who did not previously meet any of the criteria of early treatment failure;
* Presence of parasitaemia on any day between day 4 and day 28 with axillary temperature ≥ 37.5 ºC (or history of fever) in patients who did not previously meet any of the criteria of early treatment failure.

Adequate clinical and parasitological response (ACR)

- Absence of parasitemia within days 7-28 without any TF signal. For the ACR analysis, microscopic parasitological results were included with and without PCR adjustment.

Fisher's exact test was used to compare two or more independent proportions: gender, presence of symptoms, distribution of P. vivax genotype, PCR positivity and parasite persistence on days 2 and 3 between treatment groups. The Wilcoxon rank sum test was used for non-parametric comparisons: age, asexual and sexual parasitemia, drug doses, days of symptoms, and axial temperature. All tests of significance were two tailed and P values < 0.05 were considered statistically significant.

Recurrent blood infections, when detected during the 12 month follow-up were registered as well as the patients retiring. The effectiveness was calculated as the percent of the accumulated number of patients without P. vivax blood infection (first recurrent case) detected at each month of sampling, divided by the total number of patients followed up. Z test was used to determine differences in the proportion of patients or samples with a recurrent infection. To plot cumulative incidence of patient with first recurrence in percent, the Kaplan -Meier failure estimates was used.

To evaluate the clinical and parasitological outcome on primary blood infection, samples were obtained for days 2. 3, 7, 14, 21 and 28 in a flexible schedule and for recurrent blood infections were continue to sample each month up to 12 months. Blood samples from Day 2 to Day 28 were analyzed by microscopy of the thick smear and by molecular diagnosis. Samples from patient with symptoms were immediately analyzed and if a recurrent infection detected, patients were rescued by the 14-Day treatment. To uncover asymptomatic infections, all other samples within 1-12 months were analyzed by microscopy and tested antibody IgG titers and only those suspected of a recurrent blood infection were assayed by molecular diagnosis.

Only data from patients that completed the supervise treatments were include in the analysis. Parasitological and clinical cure of the primary blood infection: The analysis of response to treatment considered two outcomes based on 1) the early clinical and parasitological outcome was evaluated after 2-3 days post-treatment, 2) and therapeutic failure (TF) if clinical and/or parasitological asexual parasite persistence or reappearance occurred within 7-28 days. An adequate clinical and parasitological response (ACPR) was defined as (1) absence of parasitemia within days 7-28 without any TF signal. For the ACR analysis, microscopic parasitological results were included with and without PCR adjustment. The effectiveness for relapse elimination was evidence by the monthly follow up to one year by detecting the presence of symptoms and /or the parasite in the blood stream and the P. vivax genotype matching of primary and recurrent infections.

Classification of treatment outcomes for recurrent blood infections detected beyond 28 days and up to 12 months:

Recurrent blood infection. The recurrence of symptomatic or asymptomatic asexual parasitaemia, after or during treatment administration, can be produced by a relapse episode or a new infection. A relapse is caused by a hypnozoite, dormant stage at the liver present in s proportion of patients after a primary blood infection.

The gender, age of patients with recurrent blood infections are indicated, as well as the timing, parasitemia, serological changes , parasite genotype, presence or absence of symptoms. The proportion of recurrent episodes matching or not the genotype were compared for both treatment regimens and statistical significance calculated (p value).

SUPERVISION, FORMATS AND PROCEDURES TO AVOID MISSING DATA:

Patient registry: all documents about a patient had its name, village (and home number/ address) and the unique code. The PI was regularly supervising the procedures for diagnosis and patient recruitment and follow up at lab and field setting. The registry procedures and sheets of information per patient are kept in individual files by the PI:

* Form 1: Patient diagnosed with P. vivax: patient name, age, gender, any medication taken before diagnosis, patient address, living, asexual and sexual parasitemia per µl of blood. Name of the tutor in case it is under 18 years old patient.
* Form 2: Informed consent: one patient has met the inclusion criteria, it was asked to participate by using the informed consent of the study, approved by the ethical committee of the National Institute for Public Health in Mexico.
* Form 3: a clinical record sheet was fill in with patient´s name and unique code, clinical data from the symptomatic patient as presence of fever (within 48 h), headache, myalgias, arthralgias, symptoms suggesting paroxysm, clinical revision for the search of erythema, jaundice, and patient weight were collected.
* Form 4: follow up sheet was also implemented to register at all visits (schedule and unscheduled) the date of patient interview, clinical symptoms and blood samples collection. In case of absence of patient at home, it was annotated in the form and visit was re-schedule for the next day (in case of follow up within 28 days, but could be re-schedule within one week, or for monthly follow up (within month one to month 12).
* An Excel-data sheet data base was regularly up date (each month) and double check with the lab, field team and PI to prevent loss of information and inaccuracies.
* The slides and other samples were delivered to the laboratory wrapped in a paper with patient unique code, date of collection. Every weekday there was a reception by the same lab technician to check out all sample codes and dates with formats per patient. As the information was constantly revised, any inconsistency was resolved by samples both lab and field teams. One of two slides with thick and thin smear per time per patient were prepared and send regularly to the malaria laboratory at the National Institute for Diagnosis and Epidemiological Reference-Mexico (regularly every month), they were deliver in person by the PI as well as collection of results and any inquiry about sample´s code and results was revised and resolved. At the end of the study all samples were collected by the PI and in case of inconsistencies, samples were crossed between microscopists of the two institutions, these procedures were coordinated by the PI.

  * A copy of the follow up form was kept at the patient's home. Data checks, Source data verification to assess the accuracy: Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, etc.

The personnel involved in this project had specific tasks, and the PI regularly supervised all different activities at lab and field personnel of the study. For each patient recruited there was a schedule follow up and dates of visit programmed (one copy was provided to each patient), and when possible the cellphone of the patient or parent was useful to warn one or two prior days the next visit arrival.

Field team: comprised by two people, one clinician and one biologist. Sample reception in the Lab: was done by the same technician all over the study, separate the slides from the filter paper, and deliver and/or preserve the samples.

Microscopists: high-skilled experienced personnel, one checking samples from symptomatic patients prior to recruitment. Other microscopist was examining the slides from the study, prioritizing those samples from patients under follow up and clinically suspicious. After the examination, the slides were concentrated by the lab-supervisor and kept by the PI.

Sample size necessary to demonstrate an effect: the recommendations of the WHO for malaria treatment evaluation in the Americas were followed, but limited by the number of patients with inclusion criteria that accepted to participate during the 2 year-period. The project was also extended to nine months.

Data or samples with unclear information were discarded. They were not included in the analysis, to avoid patient lost a flexible schedule was implemented on site for missing patients Patient retirement (comprises voluntary or involuntary retirement, or protocol violation). The patient itself or patient´s tutor could retire from the study at any time, or the PI retires the patient if;

1. Presence of any concomitant disease
2. Detection of mixed Plasmodium species infection
3. Administration of other anti-malarials or extra doses of treatment during follow up
4. Patient does not wish to continue
5. Get pregnant
6. Received incomplete supervise treatment
7. Other adverse effects: severe allergies, presence of other disease by an infectious agent
8. Turn into severe malaria
9. Receiving rescue treatment

ELIGIBILITY:
Inclusion Criteria: Recommended by WHO, http://whqlibdoc.who.int/publications/2010/9789241547925_eng.pdf?ua=1

1. - Confirmed P. vivax mono- infection by microscopy
2. - Parasitemia, minimum of 500 asexual parasites per µl of blood.
3. - Presence of axillary temperature ≥ 37.5 or history of fever during the past 48 hours
4. - Ability to swallow oral medication
5. - Informed consent from the patient, or from the parent or guardian in the case of children under 7 years old, or both consents by participant and parent for individual´s age ranging within 7 and 18 years old.
6. - Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule.
7. -Patients living in accessible villages, desirable less than 1 hour far from our facility by car.

Exclusion Criteria:

1. - Mixed species infection with another plasmodium species
2. - Presence of signs of danger, or severe malaria, according to the definitions of WHO http://whqlibdoc.who.int/publications/2010/9789241547925_eng.pdf?ua=1
3. - if they presented signs of severe malnutrition or anemia
4. - had taken an anti-malaria treatment or had a malaria infection within the previous two months.
5. - Pregnant woman or positive pregnant test or breast feeding
6. - History of hypersensitivity to CQ or PQ
7. - Previous malaria attack within one year, identified at the malaria nominal record, sanitary jurisdiction VII of Chiapas, Mexico.
8. - had another cause for their fever or other chronic diseases as hypertension, diabetes, liver or kidney disease, etc.
9. - if they lived in communities at distances farther than one hour by motor vehicle from the facility.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2008-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Changes in the presence and density of asexual parasites in thick blood smears by microscopy | at days 2, 3, 7, 14, 21, 28 and monthly from month 2 to month 12, post-treatment administration
  Proportion of patients at each time-point by intervention, presenting parasitemia and mean density by examining thick blood films stained with 10% Giemsa. The two thick smears were independently examined under a light microscope using oil immersion 100 × by two trained laboratory technicians. Asexual and sexual parasite densities were determined by counting the number of parasites against 200 white blood cells (WBC) (or 500 WBC, if less than 10 parasites were encountered in 200 WBC fields), assuming 7,000 WBC/μl of blood. At least 500 fields or the whole blood smear were examined before a sample was recorded as negative.
Changes in the presence and severity of clinical symptoms | at days 2, 3, 7, 14, 21, 28 and anytime or monitor monthly during 12months, post-treatment administration
  The proportion of patients at each time-point by intervension, that present any of the following symptoms; fever, headache, myalgias, arthralgias or paroxysm were indicated by patient reference or detected by field team search; by a clinical revision of the patient, using a calibrated thermometer. Othe signs were search by the clinician as jaundice (yellowish pigmentation of the skin, the conjunctival membranes over the sclerae (whites of the eyes), erythema, herpes-like small blisters on the lips and /or outer edges of the mouth and pruritus or any itching.
Changes in the presence of recurrent infections | any time from month 1 to month 12, post T14 or during ISD treatment
  Comparing the proportion of patients presenting recurrent infections at any time schedule or unschedule (symptomatic or asymptomatic) detected by any diagnosed method

SECONDARY OUTCOMES:
Changes in the detection of parasite DNA in blood samples | at days 2, 3, 7, 14, 21, 28 and when antibody response were increased up to 12 months
  Six punches of 5 mm of dried blood in filter paper were cut and used to extract DNA using the QIAamp® DNA Blood Mini Kit, following the manufacturer instructions. To detect the P. vivax RNA ribosomal 18S subunit gene (18ssrRNA), we followed the methodology previously reported by Rubio et al. (1999).
Changes in the antibodies against blood stages of P. vivax | Monthly; from Day 28 to month 12 post-treatment administration
  Detect reduction, increases or seroconversión in the antibodies against blood stages of P. vivax per patients. From each patient, blood samples preserved in filter papers were eluted in PBS and tested in an indirect ELISA to detect IgG antibodies anti-P. vivax blood stages. The reaction was revealed using goat anti-human IgG labeled with an enzyme, and as substrate and color was recorded in a spectrophotometer. Cut off values were previously determined using unexposed individuals as the mean and 2 standard deviations; 0.25 value (95% confidence).

CONTACTS AND LOCATIONS:
Overall Officials: LILIA GONZALEZ-CERON, PHD, Principal Investigator — NATIONAL INSTITUTE FOR PUBLIC HEALTH-MEXICO

REFERENCES:
- [Background] Rodriguez MH, Betanzos-Reyes AF; Grupo de Trabajo de Malaria del Sistema Mesoamericano de Salud Publica. [Plan to improve malaria control towards its elimination in Mesoamerica]. Salud Publica Mex. 2011;53 Suppl 3:S333-48. Spanish. PMID 22344378
- [Background] White NJ. Preventing antimalarial drug resistance through combinations. Drug Resist Updat. 1998 Mar;1(1):3-9. doi: 10.1016/s1368-7646(98)80208-2. PMID 17092790
- [Background] COATNEY GR. Pitfalls in a discovery: the chronicle of chloroquine. Am J Trop Med Hyg. 1963 Mar;12:121-8. doi: 10.4269/ajtmh.1963.12.121. No abstract available. PMID 14021822
- [Background] Baird JK, Basri H, Subianto B, Fryauff DJ, McElroy PD, Leksana B, Richie TL, Masbar S, Wignall FS, Hoffman SL. Treatment of chloroquine-resistant Plasmodium vivax with chloroquine and primaquine or halofantrine. J Infect Dis. 1995 Jun;171(6):1678-82. doi: 10.1093/infdis/171.6.1678. PMID 7769318
- [Background] Galappaththy GN, Omari AA, Tharyan P. Primaquine for preventing relapses in people with Plasmodium vivax malaria. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD004389. doi: 10.1002/14651858.CD004389.pub2. PMID 17253504
- [Background] Murphy GS, Basri H, Purnomo, Andersen EM, Bangs MJ, Mount DL, Gorden J, Lal AA, Purwokusumo AR, Harjosuwarno S, et al. Vivax malaria resistant to treatment and prophylaxis with chloroquine. Lancet. 1993 Jan 9;341(8837):96-100. doi: 10.1016/0140-6736(93)92568-e. PMID 8093414
- [Background] malERA Consultative Group on Drugs. A research agenda for malaria eradication: drugs. PLoS Med. 2011 Jan 25;8(1):e1000402. doi: 10.1371/journal.pmed.1000402. PMID 21311580
- [Background] Ruebush TK 2nd, Marquino W, Zegarra J, Neyra D, Villaroel R, Avila JC, Diaz C, Beltran E. Practical aspects of in vivo antimalarial drug efficacy testing in the Americas. Am J Trop Med Hyg. 2003 Apr;68(4):391-7. PMID 12875285
- [Background] Rubio JM, Benito A, Roche J, Berzosa PJ, Garcia ML, Mico M, Edu M, Alvar J. Semi-nested, multiplex polymerase chain reaction for detection of human malaria parasites and evidence of Plasmodium vivax infection in Equatorial Guinea. Am J Trop Med Hyg. 1999 Feb;60(2):183-7. doi: 10.4269/ajtmh.1999.60.183. PMID 10072133
- [Background] Gonzalez-Ceron L, Rodriguez MH. An enzyme-linked immunosorbent assay using detergent-soluble Plasmodium vivax antigen for seroepidemiological surveys. Trans R Soc Trop Med Hyg. 1991 May-Jun;85(3):358-61. doi: 10.1016/0035-9203(91)90289-b. PMID 1949138
- [Background] Gonzalez-Ceron L, Rodriguez MH, Betanzos AF, Abadia A. [Efficacy of a rapid test to diagnose Plasmodium vivax in symptomatic patients of Chiapas, Mexico]. Salud Publica Mex. 2005 Jul-Aug;47(4):282-7. doi: 10.1590/s0036-36342005000400005. Spanish. PMID 16259289
- [Background] Gonzalez-Ceron L, Mu J, Santillan F, Joy D, Sandoval MA, Camas G, Su X, Choy EV, Torreblanca R. Molecular and epidemiological characterization of Plasmodium vivax recurrent infections in southern Mexico. Parasit Vectors. 2013 Apr 18;6:109. doi: 10.1186/1756-3305-6-109. PMID 23597046
- [Derived] Gonzalez-Ceron L, Rodriguez MH, Sandoval MA, Santillan F, Galindo-Virgen S, Betanzos AF, Rosales AF, Palomeque OL. Effectiveness of combined chloroquine and primaquine treatment in 14 days versus intermittent single dose regimen, in an open, non-randomized, clinical trial, to eliminate Plasmodium vivax in southern Mexico. Malar J. 2015 Oct 30;14:426. doi: 10.1186/s12936-015-0938-2. PMID 26518132
- See also: MEXICAN GUIDELINES THAT INCLUDE MALARIA TREATMENT NOM-032-SSA2-2002 — http://www.salud.gob.mx/unidades/cdi/nom/032ssa202.html
- See also: WHO, 2009 (METHODS FOR SURVEILLANCE OF ANTIMALARIAL DRUG EFFICACY) — http://apps.who.int/iris/bitstream/10665/44048/1/9789241597531_eng.pdf